CLINICAL TRIAL: NCT00840034
Title: A Study of Augmentation With LY2216684 for Patients With Major Depressive Disorder Who Are Partial Responders to Selective Serotonin Reuptake Inhibitor Treatment
Brief Title: A Study of Adjunctive Treatment to Antidepressant Therapy for Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12850; H9P-MC-LNDK (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-03

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2216684 (Experimental)
  Interventions: Drug: LY2216684
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2216684 — Starting dose is 6 milligrams (mg), then titrate up to 9 mg, 12 mg, or 18 mg (3 tablets) administered orally (PO), once daily (QD) for up to 10 weeks followed by a 2 week taper.
  Arms: LY2216684
Drug: Placebo — 3 tablets PO QD for up to 12 weeks
  Arms: Placebo

SUMMARY:
The primary purpose is to study the efficacy, safety, and tolerability of LY2216684 as an adjunctive treatment for participants with major depressive disorder (MDD), who were identified as partial responders to an adequate course of treatment with a selective serotonin reuptake inhibitor (SSRI) (as defined by history).

DETAILED DESCRIPTION:
This is a 12 week multi-center, double-blind, placebo-controlled study on the efficacy of LY2216684 augmentation of selective serotonin reuptake inhibitors (SSRIs) in participants with MDD who have a partial response to treatment with an SSRI. While remaining on a steady dose of their SSRI treatment at entry into the study, participants will be randomly assigned to adjunctive treatment with LY2216684 or placebo in a 1:1 ratio for 10 weeks of acute treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for major depressive disorder (MDD) as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision® (DSM-IV-TR criteria)
* Meet criteria for partial response to an adequate course of treatment defined by the investigator's opinion that participant had attained at least minimal improvement on their current Selective serotonin reuptake inhibitor (SSRI) treatment
* Women of child-bearing potential must test negative for pregnancy and agree to use a reliable method of birth control
* Grid Hamilton Rating Scale for Depression (GRID-HAMD17) total score greater than or equal 16 to at both study entry and study enrollment
* SSRI treatment for at least 6 weeks at a stable dose for at least 2 weeks prior to study enrollment
* Stated participant preference for augmentation rather than switching antidepressant treatment

Exclusion Criteria:

* Are currently involved in or discontinued within the last 30 days from a clinical trial involving an off-label use of an investigational drug
* Have previously completed or withdrawn from this study or any other study investigating LY2216684
* Have had or currently have any additional ongoing DSM-IV-TR Axis 1 condition other than MDD
* Have had any anxiety disorder preceding the onset of depression that was considered the primary diagnosis within 1 year of study entry
* Have a current or previous diagnosis of Bipolar I or II, psychotic depression, schizophrenia or other psychotic disorder
* Have a history of substance abuse within the past 1 year
* Have an Axis II disorder which, in the judgment of the investigator, would interfere with compliance with the protocol
* Have had a lack of response of the current depressive episode to 2 or more adequate courses of antidepressant therapy at a clinically appropriate dose for at least 4 weeks, or in the judgment of the investigator, the participant has treatment-resistant depression
* Have a history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), or psychosurgery within the last year
* Women who are pregnant or breastfeeding
* Participants who are judged to be at serious risk for harm to self or others
* Have a serious or unstable medical illness
* Have any diagnosed medical condition which could be exacerbated by noradrenergic agents including unstable hypertension, unstable heart disease, tachycardia or tachyarrhythmia, narrow angle glaucoma, or urinary hesitation or retention
* Have a history of severe allergies to more than 1 class of medication or multiple adverse drug reactions
* Have a history of any seizure disorder (other than febrile seizures)
* Are taking noradrenergic psychotropic medications, such as tricyclic antidepressants or serotonin norepinephrine reuptake inhibitors (SNRI)
* Have received treatment with a monoamine oxidase inhibitor (MAOI) within 14 days prior to study entry
* Require psychotropic medication other than sedative/hypnotic medication for sleep
* Are taking or have received treatment with any excluded medication within 7 days prior to study enrollment
* Have a thyroid stimulating hormone (TSH ) level outside the established reference range
* Have initiate or discontinued hormone therapy within the previous 3 months prior to enrollment
* Initiation or change in intensity of psychotherapy or other non-drug therapies within 6 weeks prior to enrollment
* A positive urine drug screen for any substance of abuse at study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- United States (24):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carson, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Costa Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Ana, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smyrna, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oak Brook, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Charles, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Willingboro, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresh Meadows, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas

REFERENCES:
- [Derived] Stauffer VL, Liu P, Goldberger C, Marangell LB, Nelson C, Gorwood P, Fava M. Is the Noradrenergic Symptom Cluster a Valid Construct in Adjunctive Treatment of Major Depressive Disorder? J Clin Psychiatry. 2017 Mar;78(3):317-323. doi: 10.4088/JCP.15m09972. PMID 27685842

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Acute Treatment Phase participants are randomized to either LY2216684 or placebo treatment groups. Participants who complete the Acute Treatment Phase or discontinue early after 4 or more weeks in the Acute Treatment phase are eligible to participate in the 2 week Taper Phase, but not all elected to participate.
Groups:
- LY2216684: LY2216684: Starting dose is 6 milligrams (mg), then titrated up to 9 mg, 12 mg, or 18 mg (3 tablets varying in strength) administered orally, once daily for up to 10 weeks, followed by a 2-week Taper Phase.
Period: Acute Treatment Phase
Arm/Group | LY2216684 | Placebo
Started | 111 | 116
Completed | 90 | 80
Not Completed | 21 | 36
Not completed — Adverse Event | 6 | 8
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 5 | 12
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 2 | 4
Not completed — Withdrawal by Subject | 6 | 11
Period: Taper Phase
Arm/Group | LY2216684 | Placebo
Started | 90 (Completed Acute Treatment (AT) or discontinued ≥4 weeks of AT and chose to participate in Taper.) | 82 (Completed Acute Treatment (AT) or discontinued ≥4 weeks of AT and chose to participate in Taper.)
Completed | 87 | 80
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- LY2216684: LY2216684: Starting dose is 6 milligrams (mg), then titrated up to 9 mg, 12 mg, or 18 mg (3 tablets, varying in strength) administered orally (PO), once daily (QD) for up to 10 weeks followed by a 2-week Taper Phase.
- Total: Total of all reporting groups
Arm/Group | LY2216684 | Placebo | Total
Number analyzed (Participants) | 111 | 116 | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (10.71) | 44.1 (10.90) | 45.0 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 79 | 158
  Male | 32 | 37 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 22 | 42
  Not Hispanic or Latino | 91 | 94 | 185
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 30 | 61
  White | 67 | 71 | 138
  More than one race | 7 | 7 | 14
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 111 | 116 | 227

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline to 8 Weeks in 16-Item Quick Inventory of Depressive Symptomatology-Self Rated (QIDS-SR16) Total Score
Description: QIDS-SR16 is a 16-item, participant-rated measure of depressive symptomatology with 4 possible answers per question that are specific to the question. Each question (Q) is scored from 0 (no problems) to 3 (increased symptoms). The total score for each visit is the sum of 9 of the 16 items: the highest number from Q1-4 (sleep), number from Q5 (feeling sad), highest number from Q6-9 (appetite and weight), total for Q10-14 (concentration, view of self, thoughts of death or suicide, general interest and energy level respectively) and the highest number from Q15-16 (psychomotor changes). The total score ranges from 0 to 27 with higher scores indicating greater severity of depression. Least Squares (LS) means are calculated using mixed model repeating measures (MMRM) and adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who do not meet response criteria during Weeks 1-2, have baseline and at least 1 post-baseline QIDS-SR16 Total Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 63 | 68
units on a scale | -4.71 (0.625) | -2.97 (0.628)

2. Secondary Outcome: Change From Baseline to 8 Weeks in 16-Item Quick Inventory of Depressive Symptomatology-Self Rated (QIDS-SR16) Individual Items
Description: QIDS-SR16 is a 16-item, participant-rated measure of depressive symptomatology with 4 possible answers per question that are specific to the question. Each question (Q) is scored from 0 (no problems) to 3 (increased symptoms). The total score for each visit is the sum of 9 of the 16 items: the highest number from Q1-4 (sleep), number from Q5 (feeling sad), highest number from Q6-9 (appetite and weight), total for Q10-14 (concentration, view of self, thoughts of death or suicide, general interest and energy level respectively) and the highest number from Q15-16 (psychomotor changes). Least Squares (LS) means are calculated using mixed model repeated measure (MMRM) and adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who do not meet response criteria during Weeks 1-2, have baseline and at least 1 post-baseline QIDS-SR16 Individual Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 63 | 68
units on a scale
  Highest Score from Items 1-4 | -0.49 (0.113) | -0.26 (0.115)
  Item 5 | -0.88 (0.124) | -0.45 (0.126)
  Highest Score from Items 6-9 | -0.32 (0.131) | -0.29 (0.133)
  Item 10 | -0.61 (0.094) | -0.33 (0.095)
  Item 11 | -0.77 (0.127) | -0.39 (0.129)
  Item 12 | -0.21 (0.048) | -0.19 (0.049)
  Item 13 | -0.55 (0.139) | -0.48 (0.140)
  Item 14 | -0.65 (0.109) | -0.28 (0.110)
  Highest Score from Items 15-16 | -0.53 (0.129) | -0.14 (0.130)

3. Primary Outcome: Change From Baseline to 8 Weeks in Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS is a 10-item checklist with items rated on a scale of 0-6, for a total scores range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) means are calculated using mixed model repeating measures (MMRM) and adjusted for investigator, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who do not meet response criteria during Weeks 1-2, have baseline and at least 1 post-baseline MADRS Total Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 62 | 68
units on a scale | -8.13 (1.251) | -5.76 (1.249)

4. Secondary Outcome: Change From Baseline to 8 Weeks in Hospital Anxiety and Depression Scale (HADS)
Description: HADS is a 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale (0-3), giving maximum scores of 21 for each subscale. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7 is 'normal.' Least Squares (LS) means are calculated using analysis of covariance (ANCOVA) and adjusted for treatment, investigator, visit, treatment-by-visit, investigator, and baseline score.
Time Frame: Baseline, up to 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who do not meet response criteria during Weeks 1-2, have baseline and at least 1 post-baseline HADS Score; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 61 | 63
units on a scale
  Anxiety Subscale Score | -2.19 (0.484) | -1.42 (0.483)
  Depression Subscale Score: number analyzed (Participants) | 61 | 62
  Depression Subscale Score | -3.28 (0.549) | -1.93 (0.551)

5. Secondary Outcome: Change From Baseline to 8 Weeks in Clinical Global Impression of Severity (CGI-S)
Description: CGI-S measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least Squares (LS) means are calculated using mixed model repeated measures (MMRM) and adjusted for treatment, investigator, visit, treatment-by visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who do not meet response criteria during Weeks 1-2, have baseline and at least 1 post-baseline CGI-Severity Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 63 | 68
units on a scale | -0.74 (0.135) | -0.71 (0.135)

6. Secondary Outcome: Change From Baseline to 8 Weeks in Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ)
Description: The CPFQ is a 7-item participant-rated questionnaire pertaining to a participant's cognitive and physical well-being. It assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each item is scored on a 6-point scale ranging from 1 (greater than normal) to 6 (totally absent). Total score ranges from 7 to 42. Higher scores indicate greater disease severity. Least Squares (LS) means are calculated using mixed model repeated measures (MMRM) and adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who do not meet response criteria during Weeks 1-2, have baseline and at least 1 post-baseline CPFQ Total Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 63 | 68
units on a scale | -5.69 (0.831) | -2.62 (0.833)

7. Secondary Outcome: Change From Baseline to 8 Weeks in Fatigue Associated With Depression Participant-Reported Outcome (FAsD PRO)
Description: The FAsD PRO is a 16-item participant-rated scale. Seven items ask how often the participants experience different aspects of fatigue with each item rated on a 5-point scale: 1 (Never) to 5 (Always). Nine items ask how often fatigue impacts various aspects of the participants lives with each item rated on a 5-point scale: 1 (Not at all) to 5 (Very much). The Fatigue Experience Score is the mean of Items 1-5, and 7, the Fatigue Impact Score is the mean of Items 8-12, 14, and 16, and the Overall Average Score is the mean of Items 1-5, 7-12, 14 and 16. The Experience, Impact and Overall Mean Scores range from 1 to 5, lower scores indicate less experience/impact. Least Squares (LS) means are calculated using analysis of covariance (ANCOVA) and adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who do not meet response criteria during Weeks 1-2, have baseline and at least 1 post-baseline FAsD-PRO Score; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 58 | 59
units on a scale
  Overall Average Score: number analyzed (Participants) | 57 | 59
  Overall Average Score | -0.75 (0.124) | -0.41 (0.127)
  Fatigue Experience Score: number analyzed (Participants) | 57 | 59
  Fatigue Experience Score | -0.60 (0.126) | -0.42 (0.129)
  Fatigue Impact Score | -0.92 (0.140) | -0.41 (0.140)

8. Secondary Outcome: Change From Baseline to 8 Weeks in Visual Analog Scale for Fatigue (VAS-F)
Description: VAS-F is a self-rated assessment on 2 items: the overall severity of fatigue and the interferences with daily activities due to fatigue. For the overall severity of fatigue the participant is asked to place a vertical mark on a 100 millimeter (mm) line between 2 anchors: 0 (not at all) and 100 (as severe as I can imagine). For the interference with daily activities due to fatigue, the participant is asked to place a vertical mark on a 100 mm line between 2 anchors: 0 (not at all) and 100 [complete disability (unable to do any activities)]. Least Squares (LS) means are calculated using analysis of covariance (ANCOVA) and adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who do not meet response criteria during Weeks 1-2, have baseline and at least 1 post-baseline VAS-F Score; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 59 | 58
units on a scale
  Severity | -16.42 (3.407) | -13.81 (3.412)
  Interference | -18.91 (3.698) | -10.33 (3.701)

9. Secondary Outcome: Change From Baseline to 8 Weeks in Visual Analog Scale for Pain (VAS-P)
Description: VAS-P is a self-rated assessment for 2 items: the overall severity of pain and the interferences with daily activities due to pain. For the overall severity of pain the participant is asked to place a vertical mark on a 100 millimeter (mm) line between 2 anchors: 0 (not at all) and 100 (as severe as I can imagine). For the interference with daily activities due to pain, the participant is asked to place a vertical mark on a 100-mm line between 2 anchors: 0 (not at all) and 100 [complete disability (unable to do any activities)]. Least Squares (LS) means are calculated using analysis of covariance (ANCOVA) and adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who do not meet response criteria during Weeks 1-2, have baseline and at least 1 post-baseline VAS-P Score; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 59 | 58
units on a scale
  Severity | -4.17 (3.450) | -0.91 (3.448)
  Interference | -9.56 (3.611) | -0.13 (3.613)

10. Secondary Outcome: Change From Baseline to 8 Weeks in Sheehan Disability Scale (SDS)
Description: The SDS is a 3-item, participant completed assessment and is used to assess the effect of the participant's symptoms on their work/social/family life. The Global Functional Impairment Total Score is a total of the 3 individual item scores, each with a scores range from 0 (not at all) to 10 (extremely). The Global Functional Impairment Total Scores range from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life. Least Squares (LS) means are calculated using analysis of covariance (ANCOVA) and adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to 8 weeks
Population: Intent-to-treat analysis is determined by treatment group participants are randomly assigned regardless of treatment received, includes all participants who do not respond in Weeks 1-2, have baseline and at least 1 post-baseline SDS Total Score; last observation carried forward. Missing work score imputed with average of other 2-item scores.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 58 | 56
units on a scale | -5.95 (1.116) | -2.63 (1.123)

11. Secondary Outcome: Change From Baseline to 8 Weeks in Quality of Life Enjoyment and Satisfaction Survey-Short Form (Q-LES-Q-SF)
Description: The Q-LES-Q-SF is a self-administered 16-item questionnaire measuring degree of enjoyment and satisfaction experienced in various areas of daily life during the past week, and is rated on a 5-point Likert scale: 1 (very poor) to 5 (very good). The Q-LES-Q-SF Total Raw Score is the sum of Items 1 to 14 and ranges from 14 to 70. The Q-LES-Q-SF Raw Scores are converted to, and expressed as the percentage of the maximum possible score. Higher scores indicate higher levels of enjoyment/satisfaction. Least Squares (LS) means are calculated using analysis of covariance (ANCOVA) and adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to 8 weeks
Population: Intent-to-treat analysis is determined by treatment group participants are randomly assigned regardless of treatment received, includes all participants who do not respond in Weeks 1-2, have baseline and at least 1 post-baseline Q-LES-Q-SF Total Score; last observation carried forward. If ≤2 items are missing mean of all other items are imputed.
Measure: Least Squares Mean (Standard Error); unit: percentage of the maximum possible score
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 59 | 58
percentage of the maximum possible score | 12.94 (2.073) | 5.44 (2.078)

12. Secondary Outcome: Change From Baseline to 8 Weeks Massachusetts General Hospital Sexual Functioning Questionnaire (MGH-SFQ)
Description: The MGH-SFQ is a 6-item participant-rated scale quantifying sexual interest, arousal (subjective excitement), ability to reach orgasm, erectile function (for males), and overall satisfaction and are scored on a 6-point scale: 1 (greater than normal) to 6 (totally absent); and overall improvement since last medication change is scored on a 6-point scale: 1 (very much improved) to 6 (much worse). Least Squares (LS) means are calculated using analysis of covariance (ANCOVA) and adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, up to 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who do not meet response criteria during Weeks 1-2, have baseline and at least 1 post-baseline MGH-SFQ Score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 103 | 104
units on a scale
  Interest | -0.70 (0.133) | -0.25 (0.136)
  Arousal | -0.74 (0.130) | -0.27 (0.132)
  Ability to Reach Orgasm | -0.81 (0.142) | -0.36 (0.144)
  Erectile Function - Males Only: number analyzed (Participants) | 31 | 31
  Erectile Function - Males Only | -0.30 (0.237) | -0.48 (0.233)
  Overall Satisfaction | -0.63 (0.141) | -0.48 (0.144)
  Overall Improvement: number analyzed (Participants) | 102 | 104
  Overall Improvement | 3.45 (0.119) | 3.62 (0.121)

13. Secondary Outcome: Colombia-Suicide Severity Rating Scale (C-SSRS)
Description: Percent of participants with suicidal ideation, behavior and acts based on C-SSRS. The C-SSRS scale captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior: a "yes" answer to any 1 of 5 suicidal behavior questions (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide). Suicidal ideation: a "yes" answer to any 1 of 5 suicidal ideation questions (wish to be dead, and 4 different categories of active suicidal ideation). Suicidal act: a "yes" answer to actual attempt or completed suicide.
Time Frame: Baseline, 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who do not meet response criteria during Weeks 1-2, have baseline and at least 1 post-baseline C-SSRS Score.
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 107 | 109
percentage of participants
  Suicidal Ideation | 11.2 | 7.3
  Suicidal Behavior | 0.9 | 0.0
  Suicidal Acts | 0.0 | 0.0

14. Other Pre Specified Outcome: Change From Baseline to 8 Weeks in Supine Systolic and Diastolic Blood Pressure
Description: Blood pressure is collected while the participant is in the supine position. Least Squares (LS) means are calculated using mixed model repeated measures (MMRM) and adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and includes all participants who have baseline and at least 1 post-baseline supine systolic and diastolic blood pressure measure.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mm Hg)
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 107 | 109
millimeters of mercury (mm Hg)
  Systolic Blood Pressure | 3.61 (1.131) | 1.31 (1.195)
  Diastolic Blood Pressure | 2.67 (0.730) | 0.77 (0.772)

15. Other Pre Specified Outcome: Change From Baseline to 8 Weeks in Supine Pulse
Description: Pulse is collected while the participant is in the supine position. Least Squares (LS) means are calculated using mixed model repeated measures (MMRM) and adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, 8 weeks
Population: Intent-to-treat population analysis is determined by the treatment groups to which participants are randomly assigned regardless of treatment received, and included all participants who have baseline and at least 1 post-baseline supine pulse rate measure.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 107 | 109
beats per minute (bpm) | 6.74 (0.986) | 0.65 (1.038)

ADVERSE EVENTS:
Groups:
- LY2216684: LY2216684: Starting dose is 6 milligrams (mg), then titrated up to 9 mg, 12 mg, or 18 mg (3 tablets, varying in strength) administered orally, once daily for up to 10 weeks followed by a 2-week Taper Phase.
- Placebo: Placebo: 3 tablets orally, once daily for up to 12 weeks.
- LY2216684-Taper Phase: LY2216684: Participants who completed or discontinued Acute Treatment Phase at or after 4 weeks were administered 12 mg orally, once daily for 1 week followed by 6 mg once daily for 1 week or 6 mg orally, once daily for 2 weeks.
- Placebo-Taper Phase: Placebo: Participants who completed or discontinued Acute Treatment Phase at or after 4 weeks continued on placebo 3 tablets orally, once daily for 2 weeks.
Arm/Group | LY2216684 | Placebo | LY2216684-Taper Phase | Placebo-Taper Phase
Serious Adverse Events (participants affected / at risk) | 3/111 | 2/116 | 1/90 | 0/82
Other Adverse Events (participants affected / at risk) | 65/111 | 48/116 | 8/90 | 8/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2216684 (N=111) | Placebo (N=116) | LY2216684-Taper Phase (N=90) | Placebo-Taper Phase (N=82)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 (N=111) | Placebo (N=116) | LY2216684-Taper Phase (N=90) | Placebo-Taper Phase (N=82)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine hypoplasia (Congenital, familial and genetic disorders) | 0/79 (0) | 1/79 (1) | 0/63 (0) | 0/59 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (8) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sluggishness (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0/79 (0) | 1/79 (1) | 0/63 (0) | 0/59 (0)
Eye burns (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (6) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Blunted affect (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatillomania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Loss of libido (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Middle insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep attacks (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Residual urine (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 1/32 (1) | 0/37 (0) | 0/27 (0) | 0/23 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 2/32 (2) | 0/37 (0) | 0/27 (0) | 0/23 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/79 (0) | 1/79 (1) | 0/63 (0) | 0/59 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 2/32 (2) | 0/37 (0) | 0/27 (0) | 0/23 (0)
Testicular swelling (Reproductive system and breast disorders) | 1/32 (1) | 0/37 (0) | 0/27 (0) | 0/23 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0/79 (0) | 1/79 (1) | 0/63 (0) | 0/59 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/79 (0) | 1/79 (1) | 0/63 (0) | 0/59 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 (8) | 1 (1) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days